CLINICAL TRIAL: NCT04168112
Title: Intracanalicular Dexamethasone Insert for Post-Corneal Cross-Linking Inflammation and Pain- The LINK Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sight Medical Doctors PLLC (Other)
Collaborators: Ocular Therapeutix, Inc. (Industry)
Responsible Party: Principal Investigator, Alanna Nattis, DO, Ophthalmologist, Director of Clinical Research, Sight Medical Doctors PLLC
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: LINK1
Record Dates: First submitted 2019-11-13; First posted 2019-11-19 (Actual); Results first posted 2024-01-30 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Keratoconus, Unstable; Collagen Crosslinking; Postoperative Pain
Keywords: Collagen Crosslinking; Keratoconus; Dexamethasone; Intracanalicular Insert
MeSH Terms: conditions — Keratoconus; Pain, Postoperative | interventions — Calcium Dobesilate; prednisolone acetate

STUDY DESIGN:
Intervention Model Description: Two cohorts of patients will be studied (10 patients each group). Cohort A: intracanalicular dexamethasone insert is placed on day of crosslinking (CXL); patients will still receive postoperative fluoroquinolone (or another class if allergy) antibiotic eye drops with instructions for use (i.e. 1 drop in operative eye 4 times daily x 10 days).
  Cohort B: Patients are placed on standard postoperative regimen of postoperative fluoroquinolone antibiotic eye drops with instructions for use (i.e. 1 drop in operative eye 4 times daily (QID) x 10 days) and Prednisolone acetate 1% ophthalmic solution tapered over 1 month in the following schedule: 4 times daily x1 week, three times daily (TID) x 1 week, twice daily (BID) x 1 week, and once daily (QD) x 1 week).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Intracanalicular dexamethasone insert is placed on day of crosslinking (CXL); patients will still receive postoperative fluoroquinolone (or other class in case of allergy) antibiotic eye drops with instructions for use (i.e. 1 drop in operative eye QID x 10 days).
  Interventions: Drug: Dextenza
- Group B (Active Comparator): Patients are placed on standard postoperative regimen of postoperative fluoroquinolone (or other class in case of allergy) antibiotic eye drops with instructions for use (i.e. 1 drop in operative eye QID x 10 days) and Prednisolone acetate 1% ophthalmic solution tapered over 1 month in the following schedule: QID x1 week, TID x 1 week, BID x 1 week, and Qday x 1 week.
  Interventions: Drug: Prednisolone Acetate

INTERVENTIONS:
Drug: Dextenza — Placement of intracanalicular dexamethasone insert for post-crosslinking inflammation and pain
  Other Names: Intracanalicular dexamethasone insert
  Arms: Group A
Drug: Prednisolone Acetate — post-crosslinking eye drop prednisolone acetate given in a tapering schedule over 1 month
  Arms: Group B

SUMMARY:
There is no standard of care medication regimen for the management of pain and inflammation post-corneal crosslinking (CXL), although most cornea specialists agree on use of an antibiotic and steroid eye drop in the immediate postoperative period. However, steroid tapering schedule and use of additional topical non-steroidal anti-inflammatory (NSAID) eyedrops vary amongst practitioners. The goal of this study is to compare postoperative pain scores between patients receiving a tapering dose of topical steroids over 1-month post-CXL, versus those receiving an intracanalicular dexamethasone insert.

DETAILED DESCRIPTION:
Keratoconus is a progressive ectatic disease of the cornea, leading to worsening of astigmatism and vision over time. With FDA approval of corneal collagen cross-linking (CXL), we now have the ability to halt the progression of keratoconus and prevent further vision loss in these patients. Although CXL has now become standard of care, the immediate post-operative period can be quite painful despite use of anti-inflammatory medications/eye drops. The goal of this study is to evaluate the efficacy of an intracanalicular dexamethasone insert in reduction of post-CXL pain as compared to routine steroid eye drop therapy.

To date, no studies have been performed evaluating the success of an intracanalicular dexamethasone insert for the treatment of postoperative inflammation and pain in corneal cross-linking patients. Oftentimes, patients experience a great deal of discomfort post-CXL, which may also make it difficult to apply eye drops in the correct fashion. Use of a dexamethasone insert alleviates the need for postoperative steroid eye drops and may provide increased pain relief post-CXL as compared to topical therapy. This will be a head-to-head study where steroid therapy (topical or insert) will begin in a standard fashion on the date of CXL. This will allow for accurate comparison of a 4-week taper of topical steroids, versus a dexamethasone insert designed to release steroid for 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Progressive keratoconus with planned corneal cross-linking in one or both eyes
* Age 18 years and older
* Ability to provide informed consent for procedures
* Ability to attend scheduled follow up visits

Exclusion Criteria:

* Age less than 18
* Pregnancy/currently breast-feeding
* Inability to provide informed consent
* Documented adverse reaction to steroid (e.g. "steroid responder", allergy, etc)
* Punctal stenosis
* Previous corneal transplant surgery
* Systemic concomitant use of controlled substance for pain management (i.e. oxycodone)
* Concurrent use of topical steroid eye drops
* Systemic, topical or intravitreal steroid use within 1 month of baseline
* Active history of chronic or recurrent inflammatory eye disease in either eye
* History of ocular herpetic infection (inclusive of Herpes Simplex 1/2, Varicella Zoster, Epstein Barr, Cytomegalovirus)
* History of neurotrophic keratitis, uncontrolled diabetes, or other disease entities that may preclude proper healing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-02-12 (Actual); Primary Completion 2022-10-24 (Actual); Study Completion 2023-04-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alanna Nattis, DO, Principal Investigator — Sight Medical Doctors PLLC
Locations (1):
- SightMD, Babylon, New York, United States

IPD SHARING:
Plan to Share IPD: No
We do not plan to share individual participant data (IPD) with other researchers. However, any adverse events will be reported to the governing institutional review board (IRB) and Ocular Therapeutix and FDA if applicable.

REFERENCES:
- [Background] Rabinowitz YS. Keratoconus. Surv Ophthalmol. 1998 Jan-Feb;42(4):297-319. doi: 10.1016/s0039-6257(97)00119-7. PMID 9493273
- [Background] Krachmer JH, Feder RS, Belin MW. Keratoconus and related noninflammatory corneal thinning disorders. Surv Ophthalmol. 1984 Jan-Feb;28(4):293-322. doi: 10.1016/0039-6257(84)90094-8. PMID 6230745
- [Background] Wollensak G, Spoerl E, Seiler T. Riboflavin/ultraviolet-a-induced collagen crosslinking for the treatment of keratoconus. Am J Ophthalmol. 2003 May;135(5):620-7. doi: 10.1016/s0002-9394(02)02220-1. PMID 12719068
- [Background] Kohlhaas M, Spoerl E, Schilde T, Unger G, Wittig C, Pillunat LE. Biomechanical evidence of the distribution of cross-links in corneas treated with riboflavin and ultraviolet A light. J Cataract Refract Surg. 2006 Feb;32(2):279-83. doi: 10.1016/j.jcrs.2005.12.092. PMID 16565005
- [Background] Hoyer A, Raiskup-Wolf F, Sporl E, Pillunat LE. [Collagen cross-linking with riboflavin and UVA light in keratoconus. Results from Dresden]. Ophthalmologe. 2009 Feb;106(2):133-40. doi: 10.1007/s00347-008-1783-2. German. PMID 18604541
- [Background] Wollensak G, Sporl E, Seiler T. [Treatment of keratoconus by collagen cross linking]. Ophthalmologe. 2003 Jan;100(1):44-9. doi: 10.1007/s00347-002-0700-3. German. PMID 12557025
- [Background] Snibson GR. Collagen cross-linking: a new treatment paradigm in corneal disease - a review. Clin Exp Ophthalmol. 2010 Mar;38(2):141-53. doi: 10.1111/j.1442-9071.2010.02228.x. PMID 20398104
- [Background] Peyman A, Kamali A, Khushabi M, Nasrollahi K, Kargar N, Taghaodi M, Razmjoo H, Fazel F, Salesi A. Collagen cross-linking effect on progressive keratoconus in patients younger than 18 years of age: A clinical trial. Adv Biomed Res. 2015 Nov 23;4:245. doi: 10.4103/2277-9175.170240. eCollection 2015. PMID 26693470
- [Background] Ghanem VC, Ghanem RC, de Oliveira R. Postoperative pain after corneal collagen cross-linking. Cornea. 2013 Jan;32(1):20-4. doi: 10.1097/ICO.0b013e31824d6fe3. PMID 22547128
- [Background] Zarei-Ghanavati S, Jafarpour S, Radyn-Majd A, Hosseinikhah-Manshadi H. Evaluation of early postoperative ocular pain after photorefractive keratectomy and corneal crosslinking. J Cataract Refract Surg. 2018 May;44(5):566-570. doi: 10.1016/j.jcrs.2018.02.019. Epub 2018 May 9. PMID 29753555
- [Background] Serna-Ojeda JC, Santana-Cruz O, Quiroz-Casian N, Gonzalez-Mendoza E, Mercado-Orozco JL, Navas A, Lichtinger A, Graue-Hernandez EO. Pain Management in Corneal Collagen Crosslinking for Keratoconus: A Comparative Case Series. J Ocul Pharmacol Ther. 2019 Jul/Aug;35(6):325-330. doi: 10.1089/jop.2019.0021. Epub 2019 Jun 19. PMID 31216215
- [Background] Kocluk Y, Cetinkaya S, Sukgen EA, Gunay M, Mete A. Comparing the effects of two different contact lenses on corneal re-epithelialization after corneal collagen cross-linking. Pak J Med Sci. 2017 May-Jun;33(3):680-685. doi: 10.12669/pjms.333.12241. PMID 28811794
- [Derived] Nattis AS, Rosenberg ED, Rasool F. Intracanalicular dexamethasone insert for post-corneal crosslinking inflammation and pain: the LINK study. J Cataract Refract Surg. 2023 Nov 1;49(11):1114-1119. doi: 10.1097/j.jcrs.0000000000001279. PMID 37532250

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Group A | Group B
Started | 10 | 10
Completed | 8 | 10
Not Completed | 2 | 0
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Population: Primary endpoints: postoperative pain between groups and degree of ocular surface inflammation.
  Secondary endpoints: rate of corneal re-epithelialization, change in intraocular pressure (mm Hg), use of rescue medications, changes in corrected distance visual acuity and central corneal pachymetry. Demographics such as age and sex were correlated with results. Notation was made of any incidence and severity of adverse events during the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A | Group B | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 10 | 20
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 26 (3.89) | 36.3 (10.29) | 31.15 (5.15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 4 | 10
  Male | 4 | 6 | 10
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: Change in Degree of Postoperative Pain Between Groups From Date of Surgery Through 1 Month Post-CXL (Day of Surgery, Postoperative Days 1 ,3, 7, Postoperative Weeks 2 ,3 and 4)
Description: Utilizing the standardized Wong-Baker visual analog pain scale, graded from 0 to 10 (no pain to increasingly worse pain (worst at 10/10))
Time Frame: Assessed at 1 day of surgery, postoperative days 1 ,3, 7, postoperative weeks 2 ,3 and 4 (7 visits total)
Population: By POD7, no patient complained of pain or discomfort (i.e, pain scale rating was "0").
Measure: Mean (Standard Deviation); unit: score on a scale from 0 - 10
Arm/Group | Group A | Group B
Number analyzed (Participants) | 8 | 10
score on a scale from 0 - 10
  Postoperative day 0 | 6.4 (1.3) | 6.6 (1.62)
  Postoperative day 1 | 1.3 (0.45) | 2 (1.18)
  Postoperative day 3 | 0.2 (0.4) | 0 (0)
  Postoperative day 7 | 0 (0) | 0 (0)
  Postoperative week 2 | 0 (0) | 0 (0)
  Postoperative week 3 | 0 (0) | 0 (0)
  Postoperative week 4 | 0 (0) | 0 (0)

2. Primary Outcome: Degree and Improvement of Ocular Surface Inflammation Between Groups From Date of Surgery Through 1 Month Post-CXL (Day of Surgery, Postoperative Days 1 ,3, 7, Postoperative Weeks 2 ,3 and 4)
Description: Assessment of corneal edema/cells (if any), degree of conjunctiva injection (if any) Grading will be from 0 to 4, with "0" being no conjunctival injection, and "4" indicating severe, diffuse conjunctival injection. Presence of corneal cells will be noted if present or absent.
Time Frame: assessed at day of surgery, postoperative days 1 ,3, 7, postoperative weeks 2 ,3 and 4 (7 visits total)
Measure: Mean (Standard Deviation); unit: score on a scale 0-4
Arm/Group | Group A | Group B
Number analyzed (Participants) | 8 | 10
score on a scale 0-4
  date of surgery | 0.5 (0) | 0.5 (0)
  postoperative day 1 | 0.5 (0) | 0.5 (0)
  postoperative day 3 | 0 (0) | 0 (0)
  postoperative day 7 | 0 (0) | 0 (0)
  postoperative week 2 | 0 (0) | 0 (0)
  postoperative week 3 | 0 (0) | 0 (0)
  postoperative week 4 | 0 (0) | 0 (0)

3. Secondary Outcome: Rate of Corneal Re-epithelialization
Description: Evaluation of rate of corneal re-epithelialization post-crosslinking at 1 day of surgery, postoperative days 1 ,3, 7, postoperative weeks 2 ,3 and 4
Time Frame: Assessed at 1 day of surgery, postoperative days 1 ,3, 7, postoperative weeks 2 ,3 and 4 (7 visits total)
Measure: Mean (Standard Deviation); unit: percentage epithelial defect
Arm/Group | Group A | Group B
Number analyzed (Participants) | 8 | 10
percentage epithelial defect
  Day of surgery | 100 (0) | 100 (0)
  Postoperative day 1 | 37.75 (5.35) | 34.75 (7.15)
  Postoperative day 3 | 7.85 (2.47) | 6 (2)
  Postoperative day 7 | 0 (0) | 0 (0)
  postoperative week 2 | 0 (0) | 0 (0)
  Postoperative week 3 | 0 (0) | 0 (0)
  Postoperative week 4 | 0 (0) | 0 (0)

4. Secondary Outcome: Subjective 'Ease of Postoperative Care' for Patients Receiving Standard Topical Steroid Eye Drop Taper vs. Dexamethasone Insert
Description: Questionnaire at final visit regarding ease of postoperative eye drop use
Time Frame: postoperative week 4 (POW4)
Population: Patients completed an ease-of-use questionnaire regarding postoperative eye drops.
Measure: Count of Participants; unit: Participants
Arm/Group | Group A | Group B
Number analyzed (Participants) | 8 | 10
Participants
  Q1. "Were directions regarding eyedrop use post-CXL easy to follow?: "yes" to Question | 8 | 10
  Q1. "Were directions regarding eyedrop use post-CXL easy to follow?: "no" to Question | 0 | 0
  Q2. "Was it cumbersome to use eyedrops for more than 10 days?": "yes" to Question | 0 | 0
  Q2. "Was it cumbersome to use eyedrops for more than 10 days?": "no" to Question | 8 | 10
  Q3. "Was it difficult to remember to use postoperative eye drops?": "yes" to Question | 0 | 0
  Q3. "Was it difficult to remember to use postoperative eye drops?": "no" to Question | 8 | 10

5. Secondary Outcome: Notation of Need for Use of "Rescue" Pain Medication
Description: Use of oral non-steroidal anti-inflammatory (NSAID), acetaminophen, prescribed pain medication) between groups
Time Frame: Assessement of use of additional/adjunctive pain/antiinflammatory medications will be done for each patient at postoperative days 1 ,3, 7, postoperative weeks 2 ,3 and 4 (7 visits total)
Population: Number of patients using "rescue" pain medication were assessed from operative day (POD0) through POW4.
Measure: Count of Participants; unit: Participants
Arm/Group | Group A | Group B
Number analyzed (Participants) | 8 | 10
Participants
  POD 0 use of pain medication | 6 | 6
  POD 1 use of pain medication | 1 | 1
  POD 3 use of pain medication | 0 | 0
  POD 7 use of pain medication | 0 | 0
  POW2 use of pain medication | 0 | 0
  POW3 use of pain medication | 0 | 0
  POW4 use of pain medication | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from baseline through the end of the study period (~1 month)
Description: The definition of adverse event/serious adverse event does not differ from clinicaltrials.gov Definitions.
Arm/Group | Group A | Group B
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/10
Other Adverse Events (participants affected / at risk) | 0/8 | 0/10

LIMITATIONS AND CAVEATS:
The biggest limitation of this study is the small sample size; 20 eyes in each group limit findings of statistical significance; larger future studies may help more definitively illuminate differences between groups. We also had 2 patients in the control group who dropped out of the study early on-data from their experiences would have been valuable in terms of comparisons between groups.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-11-20): https://cdn.clinicaltrials.gov/large-docs/12/NCT04168112/Prot_SAP_000.pdf